CLINICAL TRIAL: NCT01773837
Title: Double-blind, Placebo-controlled, Multicenter Randomized Clinical Trial to Evaluate Short-term Efficacy of Palliative Treatment With Methylphenidate in Asthenia in Advanced Cancer Patients
Brief Title: Clinical Trial to Evaluate Short-term Efficacy of Palliative Methylphenidate in Asthenia in Advanced Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual. 100 patients included
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METILAS; 2008-002171-27 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2013-01-23 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2013-08

CONDITIONS: Asthenia
Keywords: asthenia; advanced cancer; randomized controlled trial
MeSH Terms: conditions — Asthenia | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylphenidate (Experimental): methylphenidate (pill) p.o. 15 to 25 mg daily for six days
  Interventions: Drug: methylphenidate
- placebo (Placebo Comparator): the same number of pills (p.o.) than methylphenidate for six days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylphenidate — methylphenidate (pill) p.o. 15 to 25 mg daily for six days
  Arms: methylphenidate
Drug: placebo — placebo (pill) p.o.
  Arms: placebo

SUMMARY:
Fatigue is the most prevalent symptom in advanced cancer patients, interfering functional capacity, social relations, wellbeing, and quality of life. Methylphenidate is a central nervous system stimulant that has traditionally been used in cancer patients to manage depression, opioid-induced sedation, hypoactive delirium due to multiorgan failure, and cognitive disorder associated with brain tumors. Although there is evidence from prospective studies of the efficacy of this drug in cancer-related fatigue, the only one randomised clinical trials gave non-conclusive results. In order to define the real efficacy of methylphenidate in this setting, the investigators designed a new clinical trial comparing methylphenidate and placebo in cancer-related fatigue, assessed both by the verbal numeric scale (VNS) included in the Edmonton Symptom Assessment System (ESAS) and the subscale for fatigue of the Functional Assessment of Cancer Therapy (FACT-F). The investigators will include 122 advanced cancer patients with fatigue ≥ 5/10 (VNS, from 0 to 10) and hemoglobin ≥ 9 g/dl. Patients will be randomized to methylphenidate or placebo. Doses will be adapted to response within a range from 10 mg at morning time and 5 at noon, to 25 mg/day. Assessment of response will be performed on day 3 and day 6 with ESAS and FACT-F. Drug-induced adverse events will be checked. The VNS of fatigue on day 6 will be consider the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer; including metastatic, locally advanced or relapsed not amenable for curative treatment.
* Mini.mental status examination results within normal limits.
* Informed consent.
* Estimated life expectancy of at least one month.
* Hemoglobin >= 9 g/dl.
* Asthenia >= 5 (0-10; numeric verbal scale).

Exclusion Criteria:

* History of psychosis.
* Structured suicidal ideation.
* Severe anxiety.
* Severe renal, hepatic or cardiac (arrythmia, hypertension, ischemic heart disease) failure.
* Simultaneous treatment with drugs that may interact with methylphenidate as: coumarinics, anticonvulsivants (phenobarbital, phenitoin, primidone), phenylbutazone, inhibitors of mono-amine-oxidase, guanethidine.
* History of glaucoma.
* Hyperthyroidism.
* History of hypersensibility to methylphenidate.
* Clinical suspicion of: infection, hypercalcemia, hypothyroidism or renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Intensity of asthenia assessed with the verbal numeric scale (VNS) included on the Edmonton Symptom Assessment System (ESAS) | After six days of therapy
  We are looking for a difference between goups (methylphenidate versus placebo) of 1.5 (numeric rating scale: o to 10)

SECONDARY OUTCOMES:
Intensity of asthenia assessed with the subscale for fatigue of the Functional Assessment of Cancer Therapy (FACT-F) | After six days of therapy
Intensity of asthenia assessed with the verbal numeric scale (VNS) included on the Edmonton Symptom Assessment System (ESAS) and the subscale for fatigue of the Functional Assessment of Cancer Therapy (FACT-F). | After three and six days of therapy
Intensity of other symptoms assessed with the Edmonton Symptom Assessment System (ESAS) | After three and six days of treatment
Number of participants with treatment-related adverse events and severity of these adverse events. | After three and six days of treatment
  We will check for methylphenidate-related adverse events as: restlessness, hyperactivity, hyporexia, nausea and vomiting, dry mouth, palpitations, sleep insomnia, cephalea, muscle cramps, tics, and any other adverse event that could be treatment-related according to investigator. We will include the severity of the adverse event (mild, moderate, or severe), the presumed relationship with treatment, the measured required to treat it, and the final outcome.
Cognitive level. | After three and six days of treatment
  We use a specific questionnaire. In order to facilitate its use in fatigued patients it is designed with a limited number of items selected from three validated tools as MMSE, 3MS, and RBANS

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Centeno Cortes, MD, Phd, Study Chair — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided